CLINICAL TRIAL: NCT04281537
Title: A Multi-country Time and Motion Study to Describe the Experience of Clinicians, Patients and Their Caregivers During the Treatment of Fabry Disease With Enzyme Replacement Therapy With Agalsidase Alfa and Agalsidase Beta
Brief Title: A Study to Describe the Experience of Both Patients and Their Clinicians in the Treatment of Fabry Disease With Enzyme Replacement Therapy.
Status: Completed | Type: Observational
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: AT-NIS-0001
Record Dates: First submitted 2020-02-07; First posted 2020-02-24 (Actual); Results first posted 2024-11-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — Enzyme Replacement Therapy; alpha-Galactosidase; agalsidase beta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with Fabry Disease on Enzyme Replacement Therapy (ERT): Patients with Fabry Disease receiving Enzyme Replacement Therapy (agalsidase alfa or agalsidase beta)
  Interventions: Drug: Enzyme Replacement Therapy (ERT)
- Caregiver: Caregiver of patient with Fabry Disease on Enzyme Replacement Therapy (ERT)

INTERVENTIONS:
Drug: Enzyme Replacement Therapy (ERT) — ERT infusion every other week
  Other Names: agalsidase alpha; agalsidase beta
  Groups: Patient with Fabry Disease on Enzyme Replacement Therapy (ERT)

SUMMARY:
This is an international, non-interventional research study of adult patients with Fabry Disease and their caregivers. The study comprised a prospective time and motion evaluation and a cross-sectional evaluation of patient and caregiver-reported outcomes. The study evaluated the time associated with the preparation and administration of a single dose of enzyme replacement therapy (ERT) in patients by health care providers as well as the impact on Fabry patients and caregivers time and costs associated with an ERT treatment. The study also evaluated the patients' quality of life wellbeing, fatigue and work productivity.

ELIGIBILITY:
Patient Inclusion Criteria:

* Patients with a documented diagnosis of Fabry Disease (FD)
* Patients who have received ≥4 doses of ERT (with agalsidase alfa or agalsidase beta) for the treatment of FD.
* Patients who present to the participating hospital(s) or treatment centre(s) for administration of a dose of ERT (as part of their routine treatment) during the data collection period.

Caregiver Inclusion Criteria:

-Self-identifies as a caregiver of a patient with FD for whom written informed consent has been obtained for inclusion in the study.

Patient Exclusion Criteria:

* Patients who are unable or unwilling to give consent for study participation.
* Patients whose ERT preparation and administration takes place exclusively in the home setting with no healthcare professional (HCP) involvement in preparation of the infusion.
* For the time and motion evaluation: Patients whose ERT is administered by a HCP who does not consent to be observed.

Caregiver Exclusion Criteria:

- Caregiver (and/or the patient with FD whom they support or care for) is unable or unwilling to give consent for study participation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with FD who are receiving ERT and their caregivers will be identified and recruited from approximately 12 specialist centres in four countries (Taiwan, Turkey, Brazil and Japan).
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- Amicus Therapeutics, Inc., Philadelphia, Pennsylvania, United States
- Instituto de Genética e Erros Inatos do Metabolismo (IGEIM), São Paulo, Brazil
- Japan (2):
  - Keio University Hospital, Tokyo
  - Yokohama Municipal Citizen's Hospital, Yokohama
- Taiwan (2):
  - National Taiwan University, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (3):
  - Gazi University Hospital, Ankara
  - Dokuz Eylul University Medical Faculty, Izmir
  - Ege University Hospital, Izmir

REFERENCES:
- [Derived] Keyzor I, Martins AM, Ucar SK, Yamakawa H, Chien YH, Arslan N, Niu DM, Tumer L, Baldock L, Shohet S, Giuliano JD. A multi-country time and motion study to describe the experience and burden associated with the treatment of Fabry disease with enzyme replacement therapy with agalsidase alfa and agalsidase beta. Orphanet J Rare Dis. 2025 Aug 11;20(1):419. doi: 10.1186/s13023-025-03707-2. PMID 40790487

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 76 patients with Fabry Disease on enzyme replacement therapy (ERT) and 6 caregivers of patients with Fabry Disease on ERT were enrolled into the study per protocol for a total of 82 participants. As was pre-specified in the study protocol, the Agalsidase Alfa and Agalsidase Beta arms are reported as a combined group ("Patients with Fabry Disease on ERT") and not separately.
Groups:
- Patients With Fabry Disease on ERT: Patients with Fabry Disease receiving Enzyme Replacement Therapy (agalsidase alfa or agalsidase beta) infusion every other week
- Caregiver: Caregiver of patient with Fabry Disease on ERT
Period: Overall Study
Arm/Group | Patients With Fabry Disease on ERT | Caregiver
Started | 76 | 6
Completed | 76 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: As was pre-specified in the study protocol, the Agalsidase Alfa and Agalsidase Beta arms are reported as a combined group ("Patients with Fabry Disease on ERT") and not separately. Caregiver ages were reported as counts within a range.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients With Fabry Disease on ERT | Caregiver | Total
Number analyzed (Participants) | 76 | 6 | 82
Age, Continuous [Mean (Full Range); unit: years] — Population: Age of caregivers was not reported in same manner as for patients with Fabry Disease. Caregiver ages reported as counts within a range: age 31-40 (n=2), 41-50 (n=3), and 61-70 (n=1)
  years
    number analyzed (Participants) | 76 | 0 | 76
    (all) | 48.9 [19 to 74] |  | 48.9 [19 to 74]
Age, Customized [Count of Participants; unit: Participants] — Population: Caregiver ages were reported as a count within a range. Data for ages of patients with Fabry Disease on ERT are reported separately on a per patient basis
  Participants
    Caregiver age range: number analyzed (Participants) | 0 | 6 | 6
    Caregiver age range: 31 to 40 years | 0 | 2 | 2
    Caregiver age range: 41 to 50 years | 0 | 3 | 3
    Caregiver age range: 61 to 70 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 5 | 36
  Male | 45 | 1 | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 19 | 1 | 20
  Japan | 4 | 0 | 4
  Taiwan | 30 | 5 | 35
  Brazil | 23 | 0 | 23
ERT Administered to Patients [Count of Participants; unit: Participants] — Population: Type of ERT is not applicable to caregiver group
  Participants
    number analyzed (Participants) | 76 | 0 | 76
    Agalsidase alfa/biosimilar | 28 | 0 | 28
    Agalsidase beta/biosimilar | 48 | 0 | 48

OUTCOME MEASURES:

1. Primary Outcome: Total Time Spent by Healthcare Professionals (HCPs) in the Preparation/Administration of a Single Dose of ERT in Patients With Fabry Disease
Description: Total time (minutes) spent by HCPs on all activities related to administration of a single dose of ERT in patients with Fabry Disease including pre-infusion (pre-administration patient consultation; infusion and premedication preparation), ERT (and premedication) administration, and post-administration assessment and documentation. Results are shown for all patients with Fabry Disease on ERT in study
Time Frame: up to 7 weeks
Population: As was pre-specified in the study protocol, the Agalsidase Alfa and Agalsidase Beta arms are reported as a combined group ("Patients with Fabry Disease on ERT") and not separately.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Patients With Fabry Disease on ERT: Patients with Fabry Disease receiving Enzyme Replacement Therapy (ERT) (agalsidase alfa or agalsidase beta) infusion every other week
Arm/Group | Patients With Fabry Disease on ERT
Number analyzed (Participants) | 76
minutes | 151.9 (62.5)

2. Secondary Outcome: Total Time Spent by HCPs on Each Separate Task Associated With the Preparation and Administration of a Single Dose of ERT (With Agalsidase Alfa or Agalsidase Beta).
Description: Total time spent (in minutes) by healthcare professionals (HCP) on tasks associated with preparation and administration of a single dose of ERT (with agalsidase alfa or agalsidase beta) in patients with Fabry Disease including pre-administration activities (patient consultation, infusion/pre-medication preparation activities), administration of ERT (and pre-medications), and post-infusion activities (monitoring of patient during and after administration, completion of clinical documentation, and any other ERT-administration related activities).
Time Frame: up to 7 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Patients With Fabry Disease on ERT
Number analyzed (Participants) | 76
minutes
  Time Spent by HCP on Pre-infusion activities | 20.9 (13.4)
  Time spent by HCP on ERT administration | 118.2 (56.3)
  Time spent by HCP on post-infusion activities | 12.8 (9.6)

3. Secondary Outcome: Total Patient Time Associated With Attendance for the Administration of a Single Dose of ERT (With Agalsidase Alfa or Agalsidase Beta).
Description: Total patient time associated with attendance for administration of a single dose of ERT includes the total time from when the patient left home, to when they returned home and based on the reported time spent travelling, total waiting time, the total time spent during infusion episode (pre, during and post) and the other recorded activities.
Time Frame: up to 7 weeks
Population: As was pre-specified in the study protocol, the Agalsidase Alfa and Agalsidase Beta arms are reported as a combined group ("Patients with Fabry Disease on ERT") and not separately. Data were not available for 1 patient.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Patients With Fabry Disease on ERT
Number analyzed (Participants) | 75
minutes | 364.1 (193.9)

4. Secondary Outcome: Total Costs Associated With Attendance for the Administration of a Single Dose of ERT (With Agalsidase Alfa or Agalsidase Beta) - Brazil.
Description: Total out-of-pocket costs (eg, food, travel, internet) incurred by patients in Brazil that were directly related to attendance for the administration of a single dose of ERT.
Time Frame: up to 7 weeks
Population: Patients with Fabry Disease in Brazil. As was pre-specified in the study protocol, the Agalsidase Alfa and Agalsidase Beta arms are reported as a combined group ("Patients with Fabry Disease on ERT") and not separately. Data were not available for 2 patients.
Measure: Mean (Standard Deviation); unit: R$
Arm/Group | Patients With Fabry Disease on ERT
Number analyzed (Participants) | 21
R$ | 166.5 (214.8)

5. Secondary Outcome: Total Costs Associated With Attendance for the Administration of a Single Dose of ERT (With Agalsidase Alfa or Agalsidase Beta) - Taiwan.
Description: Total out-of-pocket costs (eg, food, travel, internet) incurred by patients in Taiwan that were directly related to attendance for the administration of a single dose of ERT.
Time Frame: up to 7 weeks
Population: Patients with Fabry Disease in Taiwan. As was pre-specified in the study protocol, the Agalsidase Alfa and Agalsidase Beta arms are reported as a combined group ("Patients with Fabry Disease on ERT") and not separately. Data were not available for 1 patient.
Measure: Mean (Standard Deviation); unit: NT$
Arm/Group | Patients With Fabry Disease on ERT
Number analyzed (Participants) | 29
NT$ | 709.5 (855.9)

6. Secondary Outcome: Total Costs Associated With Attendance for the Administration of a Single Dose of ERT (With Agalsidase Alfa or Agalsidase Beta) - Japan.
Description: Total out-of-pocket costs (eg, food, travel, internet) incurred by patients in Japan that were directly related to attendance for the administration of a single dose of ERT.
Time Frame: up to 7 weeks
Population: Patients with Fabry Disease in Japan. As was pre-specified in the study protocol, the Agalsidase Alfa and Agalsidase Beta arms are reported as a combined group ("Patients with Fabry Disease on ERT") and not separately.
Measure: Mean (Standard Deviation); unit: ¥
Arm/Group | Patients With Fabry Disease on ERT
Number analyzed (Participants) | 4
¥ | 8781.0 (15956.6)

7. Secondary Outcome: Total Costs Associated With Attendance for the Administration of a Single Dose of ERT (With Agalsidase Alfa or Agalsidase Beta) - Turkey
Description: Total out-of-pocket costs (eg, food, travel, internet) incurred by patients in Turkey that were directly related to attendance for the administration of a single dose of ERT.
Time Frame: up to 7 weeks
Population: Patients with Fabry Disease in Turkey. As was pre-specified in the study protocol, the Agalsidase Alfa and Agalsidase Beta arms are reported as a combined group ("Patients with Fabry Disease on ERT") and not separately. Data were not available for 1 patient.
Measure: Mean (Standard Deviation); unit: ₺
Arm/Group | Patients With Fabry Disease on ERT
Number analyzed (Participants) | 18
₺ | 470.8 (1005.5)

8. Secondary Outcome: Percentage of Patients With Work Absence Due to Attendance for This ERT Episode.
Description: The percentage of patients known to have taken time off from work during their ERT episode
Time Frame: up to 7 weeks
Population: As was pre-specified in the study protocol, the Agalsidase Alfa and Agalsidase Beta arms are reported as a combined group ("Patients with Fabry Disease on ERT") and not separately. Note: data were missing for 54% [41/76] of patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Fabry Disease on ERT
Number analyzed (Participants) | 35
Participants | 16

9. Secondary Outcome: Number of Hours of Patient Work Absence Due to Attendance for ERT Episode.
Description: The number of paid and unpaid hours that patients were absent from work during their ERT episode
Time Frame: up to 7 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Patients With Fabry Disease on ERT
Number analyzed (Participants) | 35
hours
  Number of Paid Hours Absent from Work | 6.6 (5.4)
  Number of Unpaid Hours Absent from Work | 5.3 (5.4)

10. Secondary Outcome: Total Caregiver Time Associated With Accompanying a Patient With Fabry Disease for the Administration of a Single Dose of ERT
Description: Total caregiver time (in minutes) associated with accompanying a patient with Fabry Disease for the administration of a single dose of ERT (with agalsidase alfa or agalsidase beta).
Time Frame: up to 7 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Caregiver
Number analyzed (Participants) | 6
minutes | 160 (70.43)

11. Secondary Outcome: Total Costs Associated With Accompanying a Patient With Fabry Disease for the Administration of a Single Dose of ERT
Description: Total costs associated with accompanying a patient with Fabry Disease for the administration of a single dose of ERT (with agalsidase alfa or agalsidase beta).
Time Frame: up to 7 weeks
Population: Data presented are from Taiwan in New Taiwan dollars (NT$). No data were reported for the 1 caregiver in Turkey for this outcome measure.
Measure: Mean (Standard Deviation); unit: NT$
Arm/Group | Caregiver
Number analyzed (Participants) | 5
NT$ | 2085 (1728.6)

12. Secondary Outcome: Percentage of Caregivers With Work Absence Due to Accompanying the Patient for ERT Administration.
Description: Percentage of caregivers with work absence due to accompanying the patient for this episode of ERT administration.
Time Frame: up to 7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver
Number analyzed (Participants) | 6
Participants | 3

13. Secondary Outcome: Number of Hours of Caregivers Work Absence Due to Accompanying the Patient for ERT Administration.
Description: Number of hours of caregivers work absence due to accompanying the patient for this ERT administration episode.
Time Frame: up to 7 weeks
Population: Data are available from 3 caregivers in Taiwan.
Measure: Median (Full Range); unit: hours
Groups:
- Caregiver: Caregiver of patient with Fabry Disease receiving ERT
Arm/Group | Caregiver
Number analyzed (Participants) | 3
hours
  Number of Paid Hours Absent from Work | 6.0 [6.0 to 6.0]
  Number of Unpaid Hours Absent from Work | 3.0 [1.5 to 4.5]

14. Secondary Outcome: Health Related Quality of Life (HRQoL) (12 Item Short Form Survey [SF-12] Scores / Responses)
Description: Health Related Quality of Life (HRQoL) measured by the 12 Item Short Form Survey [SF-12]). In the SF-12, patients were asked to rate aspects of their health across 8 domains; all domains have a maximum value of 5 (range 0-5) except physical functioning, for which the maximum score is 3 (range 0-3). Higher scores indicate better HRQoL while low scores indicate worse HRQoL.
Time Frame: HRQoL was completed once (during the ERT infusion visit) prior to leaving the clinic
Population: As was pre-specified in the study protocol, the Agalsidase Alfa and Agalsidase Beta arms are reported as a combined group ("Patients with Fabry Disease on ERT") and not separately. The HRQoL was completed only one time per patient.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Patients With Fabry Disease Receiving ERT: Patients with Fabry Disease receiving Enzyme Replacement Therapy (ERT) (agalsidase alfa or agalsidase beta) infusion every other week
Arm/Group | Patients With Fabry Disease Receiving ERT
Number analyzed (Participants) | 76
score on a scale
  General Health | 2.9 (1.1)
  Physical Functioning | 2.2 (0.7)
  Role Physical | 3.3 (1.1)
  Role Emotional | 3.6 (1.1)
  Bodily Pain | 3.6 (1.2)
  Mental Health | 3.5 (0.9)
  Vitality | 3.1 (1.1)
  Social Function | 3.6 (1.2)

15. Secondary Outcome: Patients General Wellbeing Measured by World Health Organization-5 Wellbeing Index (WHO-5) Scores / Responses During ERT Infusion Visit
Description: World Health Organization-5 Wellbeing Index [WHO-5] consists of 5 items and the timeframe for responses is based on the previous 2 weeks. The 5 items relate to feeling cheerful, calm, active, rested and being interested in life. For each question, patients rated the extent to which the statement applies between 0 (none of the time) and 5 (all of the time), with higher scores indicating better wellbeing. The WHO-5 total score is calculated by totaling the values of each of the five questions. The total scores range from 0 to 25, where 0 represents the worst possible quality of life and 25 represents the best possible quality of life.
Time Frame: WHO-5 was completed once (during the ERT infusion visit) prior to leaving the clinic
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Fabry Disease Receiving ERT
Number analyzed (Participants) | 76
score on a scale
  Item 1: felt cheerful and in good spirts | 3.1 (1.3)
  Item 2: felt calm and relaxed | 3.2 (1.3)
  Item 3: felt active and vigorous | 2.8 (1.4)
  Item 4: wake up feeling fresh and restful | 2.6 (1.5)
  Item 5: daily life filled with things that interest me | 3.4 (1.2)
  WHO-5 Total Score | 15.1 (5.6)

16. Secondary Outcome: Patients Level of Fatigue Measured by Fatigue Likert Scale
Description: Questionnaire measuring Fatigue. Possible scores range from 1 (not at all tired) to 5 (extremely tired); higher scores therefore indicating worse fatigue. Negative value in change from during ERT infusion to evening of ERT infusion indicates more fatigue in the evening of infusion. Negative value in change from baseline (during ERT infusion) to 1-7 days after ERT infusion indicates more fatigue during the period occurring 1-7 days after ERT infusion.
Time Frame: Questionnaire completed during ERT infusion (baseline), the same evening as date of ERT infusion, and once during the period of 1 to 7 days post-infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Fabry Disease on ERT
Number analyzed (Participants) | 76
score on a scale
  Level of fatigue during infusion | 2.4 (1.4)
  Change in level of fatigue from during ERT infusion to evening of ERT infusion | -0.2 (1.4)
  Change in level of fatigue from during ERT infusion to 1-7 days after ERT infusion | 0.1 (1.3)

17. Secondary Outcome: Patients Levels of Work Impairment (Work Productivity and Activity Index [WPAI] Scores) - 1 to 7 Days After ERT Infusion
Description: Work Productivity and Activity Index (WPAI) consists of 6 items on the effect of health problems on ability to work and perform regular activities: 1=currently employed; 2=hours missed due to health problems; 3=hours missed other reasons; 4=hours actually worked; 5=degree health affected productivity while working; 6=degree health affected regular activities
  Score calculation (multiplied by 100 for percent):
  * Percent work time missed due to health: Q2/(Q2+Q4)
  * Percent impairment while working due to health: Q5/10
  * Percent overall work impairment due to health: Q2/(Q2+Q4) + [(1-(Q2/(Q2+Q4))) x (Q5/10)]
  * Percent activity impairment due to health: Q6/10
  Final scores are expressed as impairment percentages (range: 0-100%), with higher numbers indicating greater impairment/less productivity (ie, worse outcomes) and lower numbers indicating less impairment/greater productivity (ie, better outcomes). Data were collected 1 to 7 days after ERT infusion.
Time Frame: WPAI completed once by patients during the period of 1 to 7 Days After ERT Infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Patients With Fabry Disease Receiving ERT
Number analyzed (Participants) | 76
Percent
  % Work Time Missed Due to Health (Absenteeism) | 5.0 (9.5)
  % Impairment While Working Due to Health (Presenteeism) | 28.6 (29.5)
  % Overall Work Impairment Due to Health | 28.9 (27.7)
  % Activity Impairment Due to Health | 30.8 (29.3)

18. Secondary Outcome: Patients Levels of Work Impairment (Work Productivity and Activity Index [WPAI] Scores) - Day of Next ERT Infusion
Description: Work Productivity and Activity Index (WPAI) consists of 6 items on the effect of health problems on ability to work and perform regular activities: 1=currently employed; 2=hours missed due to health problems; 3=hours missed other reasons; 4=hours actually worked; 5=degree health affected productivity while working; 6=degree health affected regular activities
  Score calculation (multiplied by 100 for percent):
  * Percent work time missed due to health: Q2/(Q2+Q4)
  * Percent impairment while working due to health: Q5/10
  * Percent overall work impairment due to health: Q2/(Q2+Q4) + [(1-(Q2/(Q2+Q4))) x (Q5/10)]
  * Percent activity impairment due to health: Q6/10
  Final scores are expressed as impairment percentages (range: 0-100%), with higher numbers indicating greater impairment/less productivity (ie, worse outcomes) and lower numbers indicating less impairment/greater productivity (ie, better outcomes). Data were collected on day of next ERT infusion.
Time Frame: WPAI completed once by patients on the day of the next ERT infusion (approximately 15 days after the prior infusion)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Patients With Fabry Disease Receiving ERT
Number analyzed (Participants) | 76
Percent
  % Work Time Missed Due to Health (Absenteeism) | 3.7 (7.3)
  % Impairment While Working Due to Health (Presenteeism) | 22.6 (24.9)
  % Overall Work Impairment Due to Health | 25.7 (26.4)
  % Activity Impairment Due to Health | 32.3 (30.4)

19. Secondary Outcome: Caregiver's Levels of Work Impairment (Work Productivity and Activity Index [WPAI]-CG Scores) - 1 to 7 Days After ERT Infusion.
Description: as for outcome 17
Time Frame: WPAI-CG completed once by caregivers during the period of 1 to 7 days after ERT infusion
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Caregiver
Number analyzed (Participants) | 6
Percent
  % Work Time Missed Due to Health (Absenteeism) | 0 (0)
  % Impairment While Working Due to Health (Presenteeism) | 17.5 (20.6)
  % Overall Work Impairment Due to Health | 17.5 (20.6)
  % Activity Impairment Due to Health | 18.3 (18.3)

20. Secondary Outcome: Caregiver's Levels of Work Impairment (Work Productivity and Activity Index [WPAI]-CG Scores) - Day of Next ERT Infusion.
Description: Work Productivity and Activity Index (WPAI) consists of 6 items on the effect of health problems on ability to work and perform regular activities: 1=currently employed; 2=hours missed due to health problems; 3=hours missed other reasons; 4=hours actually worked; 5=degree health affected productivity while working; 6=degree health affected regular activities
  Score calculation (multiplied by 100 for percent):
  * Percent work time missed due to health: Q2/(Q2+Q4)
  * Percent impairment while working due to health: Q5/10
  * Percent overall work impairment due to health: Q2/(Q2+Q4) + [(1-(Q2/(Q2+Q4))) x (Q5/10)]
  * Percent activity impairment due to health: Q6/10
  Final scores are expressed as impairment percentages (range: 0-100%), with higher numbers indicating greater impairment/less productivity (ie, worse outcomes) and lower numbers indicating less impairment/greater productivity (ie, better outcomes). WPAI was completed by caregiver on day of next ERT infusion.
Time Frame: WPAI-CG completed once by caregivers on day of the next ERT infusion (approximately 15 days after prior infusion)
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Caregiver
Number analyzed (Participants) | 6
Percent
  % Work Time Missed Due to Health (Absenteeism) | 5.0 (10.0)
  % Impairment While Working Due to Health (Presenteeism) | 17.5 (20.6)
  % Overall Work Impairment Due to Health | 21.0 (24.3)
  % Activity Impairment Due to Health | 16.7 (18.6)

21. Secondary Outcome: Level of Strain in Providing Care for a Patient With Fabry Disease (Caregiver Strain Index [CSI] Scores / Responses).
Description: The Caregiver Strain Index (CSI) consists of 12 questions with Yes/No answer and measures the strain of care provision in five domains (financial, physical, psychological, social and personal). Yes = 1 and No = 0. The range is from 0-12. Total scores are the sum of all responses. A score of 7 or higher indicates a high level of stress.
Time Frame: up to 7 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver
Number analyzed (Participants) | 6
score on a scale | 4.0 (2.3)

ADVERSE EVENTS:
Time Frame: Not applicable. Noninterventional study with no safety data collected.
Description: Not applicable. Noninterventional study with no safety data collected.
Groups:
- Patient With Fabry Disease on ERT: Patients with Fabry Disease receiving Enzyme Replacement Therapy (agalsidase alfa or agalsidase beta) infusion every other week
Arm/Group | Patient With Fabry Disease on ERT | Caregiver
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT04281537/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT04281537/SAP_001.pdf